CLINICAL TRIAL: NCT06547151
Title: A Phase 2, Prospective, Multinational, Multicenter, Double-Blind, Randomized Study to Evaluate the Safety and Efficacy of AMOR-1 as a Treatment of Hypocalcemia Associated With Hypoparathyroidism by Replacement of Currently Used Calcium Supplements (CS) in Adults.
Brief Title: Evaluating the Safety and Efficacy of AMOR-1 as a Treatment for Hypocalcemia Associated With Hypoparathyroidism in Adults
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amorphical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMCS-HP-011
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Hypoparathyroidism
Keywords: Amorphous Calcium Carbonate; hypoparathyroidism; Hypopara; Hypocalcemia; Calcium Carbonate
MeSH Terms: conditions — Hypoparathyroidism; Hypocalcemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AMOR-1 (Experimental): AMOR-1, Amorphous Calcium Carbonate (ACC) oral tablet contains 250 mg elemental calcium.
  Interventions: Drug: AMOR-1
- Active Comparator (Active Comparator): Crystalline Calcium Carbonate (CCC) oral tablet contains 500 mg elemental calcium.
  Interventions: Drug: Crystalline Calcium Carbonate

INTERVENTIONS:
Drug: AMOR-1 — Investigational arm: Tablets containing 250mg elemental calcium from Amorphous Calcium Carbonate (ACC).
  Arms: AMOR-1
Drug: Crystalline Calcium Carbonate — Control arm: Crystalline Calcium Carbonate (CCC) oral tablet contains 500 mg elemental calcium.
  Arms: Active Comparator

SUMMARY:
This clinical trial aims to evaluate the efficacy and safety of AMOR-1, consisting of Amorphous Calcium Carbonate (ACC) as the active drug substance, in treating hypocalcemia in adults with hypoparathyroidism.

DETAILED DESCRIPTION:
AMOR-1 contains Amorphous Calcium Carbonate (ACC) nanoparticles, which provide higher calcium absorption and bioavailability compared to the crystalline form. Therefore, significantly smaller doses of elemental calcium provided by ACC may be sufficient to maintain the desired serum calcium levels in people with hypoparathyroidism. The lower calcium doses can potentially reduce the adverse effects, associated with long-term, high daily doses of calcium supplementation, consumed by these patients.

The main question for the study is: Can replacing the current calcium supplement with AMOR-1, which contains half the amount of elemental calcium, maintain blood calcium levels in people with hypoparathyroidism? Patients with a history of hypoparathyroidism will be randomized in a 2:1 ratio to receive either AMOR-1 or Control (the conventional crystalline calcium carbonate supplement), respectively. Their current dose of calcium supplement will be gradually replaced with AMOR-1 or the Control over 2-4 weeks. At the end of the replacement phase, participants in the AMOR-1 arm are anticipated to receive 50% of the elemental calcium compared to their initial intake from the crystalline calcium supplements. Subjects in the Control arm will maintain their initial elemental calcium intake. Following this replacement phase, the participants will continue receiving their individual dose of AMOR-1 or the Control for an additional 10-12 weeks (Dose Maintenance phase). At the end of this phase, the participants will revert to their initial calcium supplement and will be monitored for an additional month until the end of the study. All participants will receive an active form of vitamin D in parallel to the study treatment. Throughout the study, participants will be routinely monitored for safety and efficacy, including calcium levels in the blood and urine.

ELIGIBILITY:
Inclusion Criteria:

1. An understanding, ability, and willingness to fully comply with study procedures and restrictions.
2. Ability to voluntarily provide written, signed, and dated informed consent as applicable to participants in the study.
3. Adult males or females 18 or older (prior to screening). Those < 25 years old will be examined radiologically (Bone age X-ray of non-dominant wrist and hand) to ensure epiphyseal closure prior to enrollment into the study.
4. Hypoparathyroidism patients, from any etiology, who are on currently available Standard of Care (SoC) e.g., calcium supplement and active vitamin D metabolite/analog.
5. Oral calcium ≥ 1000 mg QD above the normal dietary calcium intake
6. Albumin-adjusted total serum calcium concentration level between 7.5 mg/dL and 10.5 mg/dL, or if outside of this range, considered not clinically significant by the Investigator.
7. Vitamin D metabolite/analog therapy with calcitriol ≥0.25μg QD or alfacalcidol ≥0.50 μg QD.
8. Serum 25-hydroxyvitamin D (25OHD) ≥50 nmol/l (20 ng/ml), or if below, considered not clinically significant by the Investigator.
9. No change of treatment for hypocalcemia over the last 3 months prior to Screening as reported by the patient or through medical documentation, or if a change has occurred, it is expected to remain stable, as determined by the Investigator.
10. Absence or stable symptoms from hypocalcemia over the last 3 months prior to Screening as reported by the patient or through medical documentation.
11. For subjects receiving thyroid replacement therapy, the dose is stable for at least 6 weeks prior to screening and the TSH serum levels are within the normal range. A serum TSH level below the lower limit of the normal range but not undetectable in participant treated with thyroid hormone may be allowed if there is no anticipated need for a change in thyroid hormone dose during the trial.
12. Female subjects who are postmenopausal (12 consecutive months of spontaneous amenorrhea and age >= 51 years), or who are surgically sterilized may be enrolled, as may women of childbearing potential who had a negative pregnancy test at screening and are willing to use two medically acceptable methods of contraception for the duration of the study and undergo pregnancy testing according to the study protocol.

Exclusion Criteria:

1. Any disease that might affect calcium metabolism or calcium-phosphate homeostasis other than hypoparathyroidism, such as active hyperthyroidism, Paget's disease of bone, Type 1 or poorly controlled Type 2 diabetes mellitus (HbA1c > 9%), acromegaly, multiple endocrine neoplasia types I and II, Cushing's syndrome or disease, acute pancreatitis, malnutrition, recent prolonged immobility.
2. Severe liver disease (Child-Pugh score >9) (US FDA, 2003) or hepatic transaminases (ALT and AST) > 3 times the upper limit.
3. Severe renal insufficiency defined as estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73 m2.
4. Clinical history of symptomatic renal stones within the past 3 months. Subjects with asymptomatic renal stones are permitted.
5. Poorly controlled short bowel syndrome, bowel resection, tropical sprue, celiac disease, ulcerative colitis, and Crohn's disease.
6. Chronic or severe cardiac disease within the past 6 months including but not limited to heart failure classified as NYHA Class II-IV (Dolgin and NYHA, 1994), uncontrolled arrhythmias, bradycardia (resting heart rate < 48 beats/minute), QTc >450msec (males) or >470 msec (females) on ECG.
7. History of active or untreated malignancy (excluding thyroid cancer or basal cell skin cancer) within the past 2 years. For thyroid cancers, low-risk well-differentiated thyroid cancer that is stable does not require a disease-free period. High-risk thyroid cancer or uncontrolled cases must be disease-free for at least 1 year prior to Screening.
8. Seizure disorder/epilepsy with a history of a seizure within the previous 6 months prior to screening.
9. Acute gout within 6 months prior to screening.
10. Cerebrovascular accident within 6 months prior to Screening.
11. Subjects dependent on regular parenteral calcium infusions (e.g., calcium gluconate) to maintain calcium homeostasis.
12. Use of prohibited medications within respective prohibited periods prior to screening such as loop diuretics (30 days), raloxifene hydrochloride (3 months), lithium (30 days), methotrexate at dose >20 mg per week, or systemic corticosteroids (3 months).
13. Thiazide diuretics may be permitted if the dosage has remained stable for three months prior to screening, and there is no expected need for a dosage change during the trial.
14. Other drugs known to influence calcium and bone metabolism, such as calcitonin, cinacalcet hydrochloride, and fluoride tablets within 3 months prior to screening.
15. Use of oral bisphosphonates within 6 months or IV bisphosphonate preparations within 12 months prior to screening.
16. Previous treatment with PTH/parathyroid hormone-related protein-like drugs, including PTH(1-84) and PTH(1-34) within 30 days prior to screening.
17. Current use of Amorphous Calcium Carbonate (ACC) food supplement.
18. History of diagnosed substance abuse or alcohol dependence within the previous 3 years.
19. Pregnant/ breastfeeding patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of Subjects Who Achieved the Primary Composite Endpoint at Week 14 | 14 weeks
  The composite efficacy endpoint is defined as:
  Subject had a reduction from baseline in total daily dose of oral calcium supplementation of at least 50%, and an albumin-adjusted total serum calcium concentration level between 8.0 mg/dL (incl.) and 10.0 mg/dL (incl.), and no increase from baseline in vitamin D metabolite/analog

SECONDARY OUTCOMES:
Albumin-adjusted serum calcium | Week 4 to Week 14
  Proportion of participants who achieved albumin-adjusted serum calcium concentrations above, below, or in the range of 8.0 mg/dl and 10.0 mg/dl during Dose Maintenance.
Urinary Calcium Excretion | Week 14
  Change From Baseline in Urinary Calcium Excretion
Urine calcium excretion above 300mg/24h | Week 4 to Week 14
  Incidence of increase in urine calcium excretion (>300 mg/24h) during Dose Maintenance
GI symptoms | Week 4 to Week 14
  Incidence of GI symptoms associated with calcium intake
Symptoms associated with hypocalcemia | Week 4 to Week 14
  Incidence of symptoms associated with hypocalcemia
Hypoparathyroidism Patient Experience Scale (HPES)- Experience (HPES) - Symptom | Week 14
  Change from baseline in Hypoparathyroidism Patient Experience Scale (HPES) - Symptom total score at Week 14
HPES - Impact | Week 14
  Change from baseline in HPES - Impact total score at Week 14
HPES - Symptom - Physical Domain | Week 14
  Change from baseline HPES - Symptom - Physical Domain score at Week 14
HPES - Symptom - Cognitive Domain | Week 14
  Change from baseline in HPES - Symptom - Cognitive Domain score at Week 14
HPES - Impact - Physical Functioning Domain | eek 14
  Change from baseline in HPES - Impact - Physical Functioning Domain score at Week 14
HPES - Impact - Daily Life Domain | Week 14
  Change from baseline in HPES - Impact - Daily Life Domain score at Week 14
HPES - Impact - Psychological Well-Being Domain | Week 14
  Change from baseline in HPES - Impact - Psychological Well-Being Domain score at Week 14
HPES - Impact - Social Life and Relationships Domain | Week 14
  Change from baseline in HPES - Impact - Social Life and Relationships Domain score at Week 14
36-item Short Form (SF-36) survey | Week 14
  Change From baseline in health-related quality-of-life measured with 36-item Short Form (SF-36) survey at Week 14

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Shimon, MD, Principal Investigator — Principal Investigator
Locations (8):
- Israel (8):
  - Assuta Ashdod medical center, Ashdod, Israel
  - Hadassah Ein Kerem Medical Center, Jerusalem, Israel
  - Rabin Medical Center, Belinson Campus, Petah Tikva, Israel
  - Barzilai Medical Center, Ashkelon
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot

IPD SHARING:
Plan to Share IPD: No